CLINICAL TRIAL: NCT02086773
Title: Prospective Randomized Clinical Feasibility Study of Red Cell Transfusion Goals in Patients With Acute Leukemias
Brief Title: Red Cell Transfusion Goals in Patients With Acute Leukemias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: J13126; NA_00089706 (Other: JHM IRB)
Record Dates: First submitted 2014-03-04; First posted 2014-03-13 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Acute Promyelocytic Leukemia (APL)
Keywords: Acute Leukemia; Red Cell Transfusion
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low transfusion threshold (Experimental): Patients receive red blood cell transfusions with a transfusion threshold of 7 g/dL hemoglobin (Hb). Transfusions will not be given on schedule but will be given whenever Hb dips below the threshold.
  Interventions: Biological: Red blood cell transfusion
- High transfusion threshold (Active Comparator): Patients receive red blood cell transfusions with a transfusion threshold of 8 g/dL hemoglobin (Hb). Transfusions will not be given on schedule but will be given whenever Hb dips below the threshold.
  Interventions: Biological: Red blood cell transfusion

INTERVENTIONS:
Biological: Red blood cell transfusion
  Other Names: PRBC transfusion; RBC transfusion

SUMMARY:
The purpose of this study to determine if a lower hemoglobin transfusion threshold, 7 g/dL, has a safety profile similar to that of the current standard transfusion threshold of 8 g/dL.

DETAILED DESCRIPTION:
Transfusion of red blood cells (RBCs) is vitally important for the care of patients undergoing myelosuppressive therapy for acute leukemia. The therapeutic approach to this disease involves the use of high doses of chemotherapy to treat the blood cancers and bone marrow disorders; but it damages the marrow and blood system. Malignant and healthy stem cells are affected by the chemotherapy, and even when the malignant cells are killed, it can take weeks for the healthy cells to reconstitute the marrow. At diagnosis and before bone marrow recovery post treatment, RBCs are needed to support the patient. Current practices at major comprehensive cancer centers all utilize liberal hemoglobin transfusions triggers of 8-9 g/dL or higher. Higher hemoglobin levels in these high risk patients may have benefits such as better energy and organ function. However, research in a variety of clinical settings, suggests that a higher hemoglobin transfusion threshold is associated with the same or even higher mortality rates compared to lower hemoglobin thresholds (7-8 g/dL). These other settings include prospective randomized trials in high-risk orthopedic surgery patients, critically ill adult and pediatric ICU patients, acute GI bleed patients, and patients undergoing cardiac surgery. One clinical scenario where the ideal transfusion threshold is unknown is in patients receiving chemotherapy for hematologic malignancies. Transfusion requirements and triggers have not been systematically studied in acute leukemia or other cancers. Acute leukemia carries a high mortality; any unnecessary increase in morbidity or mortality is not acceptable. Without a clear benefit of higher transfusion thresholds, the added risks and costs of transfusion may be substantial and unnecessary. The investigators plan to study this issue in this pilot and feasibility study by randomly assigning patients treated for acute leukemia to be transfused with RBCs at either a higher or lower hemoglobin concentration trigger point. In this way, the investigators will be able to accurately determine if there is benefit or harms to having a lower or higher red cell count during the induction treatment and recovery period for patients with acute leukemias. This study will also collect information evaluating the advantages and disadvantages of the two transfusion thresholds and the feasibility of expanding the study to a large randomized trial.This safety data will serve as a platform for a larger mortality study in leukemia and possibly additional studies in solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia patients (AML, ALL, APL, treatment-related myeloid neoplasm, high grade MDS)
* Admitted with plans for inpatient myelosuppressive chemotherapy (with standard of care or protocol regimens)

Exclusion Criteria:

* Age less than 18 years
* Acute coronary syndrome as defined by active chest pain, dynamic ECG changes, troponin greater than 2.5
* Active blood loss
* Receiving erythropoietin stimulating agents prior to admission
* Chronic Renal Failure in Renal Replacement Therapy
* Documented wish against transfusion for personal or religious beliefs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Tolerance of low transfusion threshold as assessed by the percentage of participants who crossed over from the low arm to the high arm. | 60 days

SECONDARY OUTCOMES:
Safety of low vs. high transfusion threshold as assessed by total difference in number of transfusions given per participant | 60 days
  Overall safety is determined by the total difference between arms for the number of transfusions given per participant
Safety of low vs. high transfusion threshold as assessed by number of participants experiencing neutropenic infections | 60 days
  Overall safety is determined by the total difference between arms for number of participants experiencing neutropenic infections, where neutropenia is defined as absolute neutrophil count < 500/mcL.
Safety of low vs. high transfusion threshold as assessed by number of grade 3-4 bleeding events as defined by CTCAE 4.0 | 60 days
Safety of low vs. high transfusion threshold as assessed by number of deaths attributed to induction chemotherapy | 60 days
Safety of low vs. high transfusion threshold as assessed by number of participants with at least one grade 3-5 non-hematological toxicity by CTCAE 4.0. | 60 days
Feasibility as determined by percentage of participants consented | 60 days
  As per protocol-defined criteria, the transfusion strategy being tested would be deemed feasible if all of the following criteria are met: 1) More than 50% of eligible patients could be consented; 2) More than 75% of participants randomized to the low arm tolerated the 7 g/dL transfusion threshold; 3) Fewer than 15% of participants crossed over from the low arm to the high arm; 4) The study was not paused for safety concerns.
Feasibility as determined by percentage of participants who tolerate 7g/dL transfusion | 60 days
  As per protocol-defined criteria, the transfusion strategy being tested would be deemed feasible if all of the following criteria are met: 1) More than 50% of eligible patients could be consented; 2) More than 75% of participants randomized to the low arm tolerated the 7 g/dL transfusion threshold; 3) Fewer than 15% of participants crossed over from the low arm to the high arm; 4) The study was not paused for safety concerns.
Feasibility as determined by percentage of participants who crossed over from the low arm to the high arm | 60 days
  As per protocol-defined criteria, the transfusion strategy being tested would be deemed feasible if all of the following criteria are met: 1) More than 50% of eligible patients could be consented; 2) More than 75% of participants randomized to the low arm tolerated the 7 g/dL transfusion threshold; 3) Fewer than 15% of participants crossed over from the low arm to the high arm; 4) The study was not paused for safety concerns.
Number of transfusions | 60 days
  Median number of red cell and platelet transfusions given per participant.
Neutropenic infections | 60 days
  Number of participants in each arm experiencing neutropenic infections, where neutropenia is defined as absolute neutrophil count < 500/mcL.
Bleeding | 60 days
  Number of grade 3-4 bleeding events as defined by CTCAE 4.0.
Length of stay | 60 days
  Median length of inpatient stay in days. This is for the initial inpatient stay for induction chemotherapy only (chemotherapy itself was not part of this protocol).
Treatment-related mortality | 60 days
  Number of deaths attributed to induction chemotherapy.
End organ dysfunction | 60 days
  Number of participants with at least one grade 3-5 nonhematological toxicity as defined by CTCAE 4.0.
Performance status scores | 60 days
  Number of participants with Eastern Cooperative Oncology Group (ECOG) performance status < 2. The ECOG scale is rated from 0 to 5, where 0 is best health and 5 is dead.
Incidence of crossover | 60 days
  Number of participants who crossed over from the low to the high arm due to symptomatic anemia (defined as Hb < 8 g/dL with symptoms).
Cost savings | 60 days
  Estimated per-patient cost savings of the low transfusion threshold compared to the high transfusion threshold.
Fatigue scores | 60 days
  Median difference in fatigue scores as graded on the National Cancer Institute Fatigue Scale. Scores are from 0 to 10, where 0 is no fatigue and 10 is the worst possible fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Amy DeZern, MD, MHS, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DeZern AE, Williams K, Zahurak M, Hand W, Stephens RS, King KE, Frank SM, Ness PM. Red blood cell transfusion triggers in acute leukemia: a randomized pilot study. Transfusion. 2016 Jul;56(7):1750-7. doi: 10.1111/trf.13658. Epub 2016 May 20. PMID 27198129
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836